CLINICAL TRIAL: NCT04294199
Title: Effect of Early Range of Motion on Recovery in Individuals Following First Time Patellar
Brief Title: Effect of Early Range of Motion Following First Time Patellar Dislocation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Scott McKay, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H43929
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Patellar Dislocation
MeSH Terms: conditions — Patellar Dislocation | interventions — Immobilization

STUDY DESIGN:
Intervention Model Description: Dual-arm randomized intervention comparison study evaluation two rehabilitation protocols for individuals following a first time lateral patella instability episode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immobilization (Active Comparator): Patients in this group will be given a knee immobilizer to wear for 2 weeks and then receive outpatient physical therapy evaluation and treatment
  Interventions: Other: Early Range of MOtion
- Early range of motion (Experimental): Patients in this group will be allowed to move the knee and start outpatient physical therapy and treatment immediately.
  Interventions: Other: Early Range of MOtion

INTERVENTIONS:
Other: Early Range of MOtion — Groups will be compared to see if immobilization or early range of motion is better at returning to their sport after patellar dislocation.
  Other Names: Immobilization; Ear;y Range of Motion

SUMMARY:
Do teen-age patients with a dislocated knee cap do better with or without a brace?

DETAILED DESCRIPTION:
This study will look at two different ways to treat teen-age patients who have had a dislocation of their knee cap. Both groups will receive the physical therapy treatment for knee cap dislocation but one group will first be in a brace for a week and the other group will start moving in therapy right away.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents between 11-17 years
* Medical diagnosis of 1st time lateral patellar instability episode (dislocation or subluxation)
* Subjective history of knee shifting, instability, popping out, knee effusion
* Apprehension test is positive and has medial patellar tenderness
* Referred to the Texas Children's Hospital (TCH) outpatient sports medicine clinic from an emergency room facility, urgent care or pediatrician within 10 days of the injury.
* Free of co-morbidities that would prevent or limit rehabilitation including cardiac, pulmonary, psychiatric (except Attention Deficit Disorder (ADD) or Attention Deficit Hyperactivity Disorder (ADHD), orthopedic, neurological
* Must be able to follow directions and participate in rehabilitation protocol for the 3-month study period.

Exclusion Criteria:

* Imaging or clinical findings suggest surgical intervention is needed i.e. fracture, osteochondral defect, Lachman or other positive knee ligament special tests.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-10-31 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Kujala Knee Score | 10 minutes
  13 item questionnaire to rate pain, function, ambulation, and instability
Tegner Activity Scale | 5 minutes
  11 levels of activity from complete inability to function to advanced sports participation
Isokinetic Strength using Biodex | 30 minutes
  Force of movement is measured in newtons and torque and corrected for body weight
Passive Range of Motion | 5 minutes
  Measured with goniometer to record full range of motion in knee flexion and extension
Edema Assessment | 2 minutes
  Measure of knee circumference

SECONDARY OUTCOMES:
Numerical Pain Rating Scale | 1 minute
  Pain rated by patient on scale of 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Scott McKay, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erickson BJ, Mascarenhas R, Sayegh ET, Saltzman B, Verma NN, Bush-Joseph CA, Cole BJ, Bach BR Jr. Does Operative Treatment of First-Time Patellar Dislocations Lead to Increased Patellofemoral Stability? A Systematic Review of Overlapping Meta-analyses. Arthroscopy. 2015 Jun;31(6):1207-15. doi: 10.1016/j.arthro.2014.11.040. Epub 2015 Jan 28. PMID 25636989
- [Result] Armstrong BM, Hall M, Crawfurd E, Smith TO. A feasibility study for a pragmatic randomised controlled trial comparing cast immobilisation versus no immobilisation for patients following first-time patellar dislocation. Knee. 2012 Oct;19(5):696-702. doi: 10.1016/j.knee.2011.08.004. Epub 2011 Sep 29. PMID 21962458
- [Result] Saccomanno MF, Sircana G, Fodale M, Donati F, Milano G. Surgical versus conservative treatment of primary patellar dislocation. A systematic review and meta-analysis. Int Orthop. 2016 Nov;40(11):2277-2287. doi: 10.1007/s00264-015-2856-x. Epub 2015 Jul 23. PMID 26202017
- [Result] Cheng B, Wu X, Ge H, Qing Sun Y, Zhang Q. Operative versus conservative treatment for patellar dislocation: a meta-analysis of 7 randomized controlled trials. Diagn Pathol. 2014 Mar 18;9:60. doi: 10.1186/1746-1596-9-60. PMID 24636710
- [Result] Matic GT, Magnussen RA, Kolovich GP, Flanigan DC. Return to activity after medial patellofemoral ligament repair or reconstruction. Arthroscopy. 2014 Aug;30(8):1018-25. doi: 10.1016/j.arthro.2014.02.044. Epub 2014 Apr 24. PMID 24768468
- [Result] Vavken P, Wimmer MD, Camathias C, Quidde J, Valderrabano V, Pagenstert G. Treating patella instability in skeletally immature patients. Arthroscopy. 2013 Aug;29(8):1410-22. doi: 10.1016/j.arthro.2013.03.075. Epub 2013 May 25. PMID 23714402